CLINICAL TRIAL: NCT06045442
Title: Exercise During Hemodialysis With a Bed Compatible Trainingstool: a Randomized Controlled Trial
Brief Title: Dialysis Exercise With a Bed Compatible Leg TRAiningstool
Acronym: DEXTRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-40-B
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Chronic Kidney Diseases; Hemodialysis
Keywords: Dialysis; Intradialytic exercise; Hemodialysis training
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Random assignment in 1:1 ratio to either the intervention group (intradialytic exercise; twice a week for 30 min per dialysis session) or control group (Usual care)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 3 months intradialytic exercise intervention: 30 minutes of endurance training at the dialysis unit with a dialysis training device, twice a week.
  Interventions: Behavioral: Intradialytic exercise training
- Control (Active Comparator): Usual Care
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Intradialytic exercise training — The patients in the intervention group will receive 3 months of endurance training, 2x/week for 30 min. 5 min of this should be a warm-up, 20 min of exertion and 5 min of cool down. The warm-up and cool-down should be equivalent to a very light load (Borg scale 9), whereas the exertion phase should be exhausting for the patients (Borg scale 14-15).
  Arms: Intervention
Behavioral: Control — Usual care
  Arms: Control

SUMMARY:
This study is a randomised controlled intervention trial for dialysis patients with chronic kidney disease (n=32). The aim of this study is to test the effectiveness of an intradialytic training with a simple bed compatible trainingstool in comparison to a control group.

DETAILED DESCRIPTION:
Patients are randomised to either the intervention or control group at the beginning of the study. Both groups are evaluated at the beginning and after 2 months regarding their body composition, physical performance, fatigue and quality of life. The control group receives usual care. The intervention group receives an intradialytic exercise training with a bed compatible trainingstool.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years
* Patients who started dialysis more than 3 months ago
* Patients must be mentally and physically able to participate in exercise

Exclusion Criteria:

* Patients who are not mentally or physically able to participate in intradialytic exercise. These include patients with uncontrolled high blood pressure and uncontrolled diabetes mellitus, diseases that impair physical performance or/and could be aggravated by activity, such as ischaemic cardiopathy or symptoms associated with coronary heart disease, chronic coronary heart disease, chronic lung disease and orthopaedic conditions that make exercise impossible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
Sit-to-stand test (STS60) | 3 month
  measured in number of repetitions in 60 seconds
Timed-up-and-go test (TUG) | 3 month
  measured in time (seconds)

SECONDARY OUTCOMES:
muscle mass | 3 month
  measured in kg by bio-impedance analysis
body fat mass | 3 month
  measured in kg by bio-impedance analysis
Quality of life by Kidney Disease Quality of Life Instrument (KDQOL) | 3 month
  measured in change of scale by questionnaire (higher Score = better health; Questions are combined to form items and the average is calculated; Range from 0-100)
Fatigue by Fatigue Assessment Scale (FAS) | 3 month
  measured in change of scale by questionnaire (scores can range from 10 (lowest level of fatigue) to 50 (highest level of fatigue)
activity by Freiburg Questionnaire of physical activity | 3 month
  measured in change of scale by questionnaire (The higher the score, the more active the participant. the lowest level would be a score of 0)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Schiffer, Prof., Study Director — Universitätsklinikum Erlangen
Locations (1):
- Universitätsklinikum Erlangen, Erlangen, Bavaria, Germany